CLINICAL TRIAL: NCT03995615
Title: To Estimate the Levels of Gingival Crevicular Fluid YKL-40 in Patients With Healthy Periodontium, Chronic Periodontitis and Chronic Periodontitis With Rheumatoid Arthritis Following Scaling and Root Planing A Clinico-biochemical Study
Brief Title: ESTIMATION OF GINGIVAL CREVICULAR LEVEL OF YKL40
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, professor/ head of the department periodontology, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_91499
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Periodontitis and Rheumatoid Arthritis
MeSH Terms: conditions — Periodontitis; Arthritis, Rheumatoid | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: * Group I (Control) - 15 periodontally healthy patient with probing depth< 3mm
  * Group II - 15 systemically healthy chronic periodontitis patient who had >25% of sites with gingival bleeding and an absence of probing depth ≥ 4mm and clinical attachment level ≥3mm
  * Group III - 15 chronic periodontitis patient with a probing depth ≥ 5mm and relative attachment loss of ≥8mm and ≥ 10% sites with bleeding on probing present with radiographic evidence of bone loss and Rheumatoid arthritis with diseases active score 28[DAS-28] ≥3.2 to ≤5.1with out scaling and root planing.
  * Group IV - 15 chronic periodontitis patient with a probing depth ≥ 5mm and relative attachment loss of ≥8mm and ≥ 10% sites with bleeding on probing present with radiographic evidence of bone loss and Rheumatoid arthritis with diseases active score 28[DAS-28] ≥3.2 to ≤5.1 with scaling and root planing. Periodontal clinical parameters will be assessed.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group I (Control) (No Intervention): • Group I (Control) - 15 periodontally healthy patient with probing depth< 3mm and ≤ 10% sites with bleeding on probing.
- • Group II (No Intervention): • Group II - 15 systemically healthy chronic periodontitis patient who had presented >25% of sites with gingival bleeding ,surface demonstrating supra-gingival plaque accumulation and an absence of probing depth ≥ 4mm and clinical attachment level ≥3mm
- • Group III (No Intervention): • Group III - 15 chronic periodontitis patient with a probing depth ≥ 5mm and relative attachment loss of ≥8mm and ≥ 10% sites with bleeding on probing present with radiographic evidence of bone loss and Rheumatoid arthritis with diseases active score 28[DAS-28] ≥3.2 to ≤5.1with out scaling and root planing
- • Group IV (Active Comparator): • Group IV - 15 chronic periodontitis patient with a probing depth ≥ 5mm and relative attachment loss of ≥8mm and ≥ 10% sites with bleeding on probing present with radiographic evidence of bone loss and Rheumatoid arthritis with diseases active score 28[DAS-28] ≥3.2 to ≤5.1 with scaling and root planing. Periodontal clinical parameters will be assessed
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Procedure: scaling and root planing — * After initial clinical evaluation, supra gingival calculus removal will be done. GCF samples will be collected from the control and test groups (Baseline samples) using paper strips (ORAFLOW). ® Group III patients will undergo a through oral hygiene instructions, full mouth supra-gingival and sub- gingival scaling and root planing clinical parameters will be re-recorded 6 weeks later and a 2nd GCF samples will be collected from selected test site from each patients following periodontal intervention.
  * All the samples will be placed in eppendorf vials containing the buffer solution and samples will be stored at -800 c until the time of analysis by Enzyme -linked immune sorbent assay kit (ELISA) (GENX BIO) TM
  Arms: • Group IV

SUMMARY:
The presence of YKL- 40 an acute phase protein in both chronic periodontitis and rheumatoid arthritis. However, till date no studies has been done on the levels of gingival crevicular fluid YKL-40 following scaling and root planing, the present study which is first of its kind is designed to detect and estimate the gingival crevicular fluid YKL-40 levels in healthy patients, chronic periodontitis and patient with chronic periodontitis having rheumatoid arthritis at baseline and chronic periodontitis having rheumatoid arthritis 6 weeks post periodontal therapy (scaling and root planning [SRP]). This could throw more light on it and extend our knowledge on its role in both the conditions.

DETAILED DESCRIPTION:
Periodontal diseases is a chronic inflammatory diseases initiated by microbial infection that leads to a host response resulting in inflammatory breakdown of tooth supporting, osseous and soft tissue structures YKL-40 also called as human cartilage glycoprotein-39(HC-gp39), an acute phase protein is a novel potential bio marker in relation to both acute and chronic inflammations. YKL-40 is a member of "mammalian chitinase- like protein" but has no chitinase/ enzymatic activity, with molecular weight of approximately 40KDa. It is named from three amino acids of Tyrosine (Y), Lysine (K) and leucin (L) at the N-terminal YKL-40 was identified in gingival crevicular fluid (GCF) and serum among gingivitis and periodontitis individual with or without diabetic mellitus. Investigation was done in association between chronic periodontitis and diabetic mellitus in gingival crevicular fluid sample. However, the past studies have reported an increased prevalence of rheumatoid arthritis in patient with periodontal diseases. They have reported the presence of rheumatoid factor in gingiva, sub gingival plaque, saliva and serum of periodontally diseased patient. Treatment of periodontal disease has demonstrated significant reduction in erythrocyte sedimentation rate (ESR) which in turn have showed improvement of clinical indices on rheumatoid arthritis activity.we speculate that presence of YKL 40 an acute phase protein in both chronic periodontitis and rheumatoid arthritis. However, till date no studies has been done on the levels of gingival crevicular fluid YKL-40 following scaling and root planing, the present study which is first of its kind is designed to detect and estimate the gingival crevicular fluid YKL-40 levels in healthy patients, chronic periodontitis and patient with chronic periodontitis having rheumatoid arthritis at baseline and chronic periodontitis having rheumatoid arthritis 6 weeks post periodontal therapy (scaling and root planning [SRP]). This could throw more light on it and extend our knowledge on its role in both the condition

ELIGIBILITY:
Inclusion Criteria:

* 1. Age group of 25 to 55 years. 2. Patient diagnosed with active rheumatoid arthritis with DAS scoring between ≥3.2 to ≤5.1 3. Patient with generalized mild to moderate chronic periodontitis. 4. Patient who had not received any periodontal treatment in last six months. 5. Dentition with at least twenty functioning teeth. 6. Patient who are co-operative and able to attend follow-up.

Exclusion Criteria:

* 1. Any systemic diseased such as diabetic mellitus and thyroid diseases. 2. Former and current smokers. 3. Pregnant and lactating females. 4. Usage of antibiotics or patients on Diseases Modifying Anti-Rheumatic Drugs (DMARD) that affects the periodontal status in the last six months.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
levels of YKL40 IN GCF | 6 WEEEKS
  To estimate the levels of gingival crevicular fluid YKL-40 in patients with healthy periodontium, chronic periodontitis and chronic periodontitis with rheumatoid arthritis following scaling and root planing

CONTACTS AND LOCATIONS:
Overall Officials: RUDRAKSHI C, MDS, Principal Investigator — Krishnadevaraya college of dental sciences , Banglore ,KARNATAKA , INDIA
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
IPD are personal informations of patients and its confidential .